CLINICAL TRIAL: NCT02451943
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial of Doxorubicin Plus Olaratumab Versus Doxorubicin Plus Placebo in Patients With Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: A Study of Doxorubicin Plus Olaratumab (LY3012207) in Participants With Advanced or Metastatic Soft Tissue Sarcoma
Acronym: ANNOUNCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15677; I5B-MC-JGDJ (Other: Eli Lilly and Company); 2015-000134-30 (EudraCT Number)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Soft Tissue Sarcoma
Keywords: leiomyosarcoma; soft tissue sarcoma (STS); advanced soft tissue sarcoma; metastatic soft tissue sarcoma; liposarcoma; undifferentiated pleomorphic sarcoma; doxorubicin
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma; Liposarcoma; Histiocytoma, Malignant Fibrous | interventions — olaratumab; Doxorubicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxorubicin + Olaratumab (Experimental): 75 milligrams per meter squared (mg/m^2) doxorubicin administered intravenously (IV) on day 1 of each 21-day cycle for 8 cycles plus 20 milligrams per kilogram (mg/kg) dose of olaratumab administered IV on day 1 and day 8 of cycle 1 and 15 mg/kg olaratumab administered IV on day 1 and day 8 of cycles 2-8. Beginning with cycle 9, 15 mg/kg olaratumab administered IV on day 1 and day 8 of each subsequent 21-day cycle until documented progressive disease (PD) or discontinuation for any other reason.
  Interventions: Drug: Olaratumab; Drug: Doxorubicin
- Doxorubicin + Placebo (Placebo Comparator): 75 mg/m^2 doxorubicin administered IV on day 1 of each 21-day cycle for 8 cycles plus placebo (equivalent volume) administered IV on day 1 and day 8 for 8 cycles. Beginning with cycle 9, placebo (equivalent volume) administered on days 1 and 8 of each subsequent 21-day cycle until PD or discontinuation for any other reason.
  Interventions: Drug: Doxorubicin; Drug: Placebo

INTERVENTIONS:
Drug: Olaratumab — Administered IV
  Other Names: LY3012207
  Arms: Doxorubicin + Olaratumab
Drug: Doxorubicin — Administered IV
Drug: Placebo — Administered IV
  Arms: Doxorubicin + Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of the combination of doxorubicin plus the study drug known as olaratumab versus doxorubicin plus placebo in participants with advanced or metastatic soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced unresectable or metastatic soft tissue sarcoma not amenable to curative treatment with surgery or radiotherapy. Participants with Kaposi's sarcoma and gastrointestinal stromal tumors (GIST) will be excluded. Note: Evidence of disease progression is required for participants that are not newly diagnosed.
* Presence of measurable or nonmeasurable but evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1, Eisenhauer et al. 2009).
* Performance status 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* The participant has not received any previous treatment with anthracyclines.
* The participant may have had any number of prior systemic cytotoxic therapies for advanced/metastatic disease and are considered appropriate candidates for anthracycline therapy. All previous anticancer treatments must be completed ≥ 3 weeks (21 days) prior to first dose of study drug.
* Availability of tumor tissue is required for study eligibility. The participant must have consented to provide archived formalin-fixed paraffin embedded (FFPE) tumor tissue or be subject to a pre-treatment re-biopsy of primary or metastatic tumor tissue for future central pathology review and translational research (if archived tissue is unavailable).
* Adequate hematologic, organ, and coagulation within 2 weeks (14 days) prior to randomization.
* Left ventricular ejection fraction (LVEF) ≥50% assessed within 28 days prior to randomization.
* Females of child-bearing potential must have a negative serum pregnancy test within 7 days prior to randomization.
* Females of child-bearing potential and males must agree to use highly effective contraceptive precautions during the trial and up to 3 months following the last dose of study drug.
* The participant has, in the opinion of the investigator, a life expectancy of at least 3 months.

Exclusion Criteria:

* Diagnosis of GIST or Kaposi sarcoma.
* Active central nervous system (CNS) or leptomeningeal metastasis (brain metastasis) at the time of randomization. Participants with a history of a CNS metastasis previously treated with curative intent (for example, stereotactic radiation or surgery) that have not progressed on follow-up imaging, have been asymptomatic for at least 60 days and are not receiving systemic corticosteroids and or/anticonvulsants, are eligible. Participants with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before randomization to rule out brain metastasis.
* Prior treatment with doxorubicin, epirubicin, idarubicin, and/or other anthracyclines or anthracenediones; the participant has received treatment with olaratumab or has participated in a prior olaratumab trial.
* Prior radiotherapy of the mediastinal/pericardial area or whole pelvis radiation.
* The participant has symptomatic congestive heart failure (CHF), left ventricular dysfunction (LVEF < 50%), severe myocardial insufficiency, cardiac arrhythmia, or cardiomyopathy.
* The participant has unstable angina pectoris, angioplasty, cardiac stenting, or myocardial infarction within 6 months of randomization.
* The participant has a QT interval calculated using Bazett's formula (QTcB) interval of >450 milliseconds (msec) for males and >470 msec for females on screening electrocardiogram (ECG).
* Females who are pregnant or breastfeeding.
* Known allergy to any of the treatment components including a history of allergic reactions attributed to compounds of chemical or biological composition similar to olaratumab.
* The participant has a known active fungal, bacterial, or viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (111):
- United States (27):
  - City of Hope National Medical Center, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Georgia Cancer Specialists PC, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University Medical School, St Louis, Missouri
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Oncology Hematology Care Inc, Fairfield, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The West Clinic, Germantown, Tennessee
  - Oncology Hematology Care Inc, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Fairfax Northern Virginia Hematology Oncology, PC, Fairfax, Virginia
- Argentina (3):
  - Alexander Fleming, CABA, BS
  - CENIT Centro de Neurociencias, Investigación y Tratamiento, Caba, Buenos Aires
  - Hospital Provincial del Centenario, Rosario, Santa Fe Province
- Chris O'Brien Lifehouse, Camperdown, New South Wales, Australia
- AKH, Vienna, Austria
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels, Brussels Capital
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Brazil (2):
  - INCA Hospital do Câncer III, Rio de Janeiro, Rio de Janeiro
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo, São Paulo
- Canada (4):
  - Tom Baker Cancer Center, Calgary, Alberta
  - BC Cancer Vancouver, Vancouver, British Columbia
  - Princess Margaret Hospital (Ontario), Lai Chi Kok, Kowloon
  - Royal Victoria Hospital-Montreal, Montreal, Quebec
- Herlev and Gentofte Hospital, Herlev, Denmark
- Finland (2):
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Turku University Central Hospital, Turku
- France (7):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - CHU Hopital d'enfants de la Timone, Marseille
  - Institut Curie, Paris
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (5):
  - Klinikum Mannheim gGmbH Universitätsmedizin, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Klinikum der Universität München Großhadern, München, Bavaria
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - HELIOS Klinikum Berlin-Buch, Berlin
- Magyar Honvedseg Egeszsegugyi Kozpont, Budapest, Hungary
- Israel (3):
  - Sheba Medical Center, Tel Litwinsky, Ramat Gan
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Istituto Nazionale dei Tumori, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Università degli Studi di Catania - Azienda Policlinico, Catania, Sicily
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
- Japan (11):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Osaka University Hospital, Suita, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Okayama University Hospital, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
- Mexico (5):
  - Hospital Angeles, Tijuana, Estado de Baja California
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Consultorio Dr. Reinoso, Monterrey, Nuevo León
  - Centro de Atención E Investigación Clínica En Oncología, Mérida, Yucatán
  - Centro de Alta Especialidad Reumatologia Inv del Potosi SC, San Luis Potosí City
- Netherlands (5):
  - Maastricht UMC+, Maastricht, Limburg
  - University Medical Center Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Universitair Medisch Centrum St Radboud Nijmegen, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw, Poland
- Russia (3):
  - Kazan Oncology Dispensary, Kazan', Tatarstan Republic
  - Blokhin Cancer Research Center, Moscow
  - St-Petersburg scientifical practical cente spec medical care, Saint Petersburg
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Asan Medical Center, Seoul, Korea
  - Seoul St. Mary's Hospital, Seoul, Korea
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Universitario Virgen Del Rocio, Seville, Andalusia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Duran I Reynals, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Fe de Valencia, Valencia
- Skånes universitetssjukhus Lund, Lund, Sweden
- Switzerland (2):
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - Inselspital Bern, Bern
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan Hsien
- United Kingdom (5):
  - University College Hospital - London, London, Greater London
  - Royal Marsden NHS Trust, London, Greater London
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - The Clatterbridge Cancer Centre, Bebbington, Merseyside
  - Weston Park Hospital, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Jones RL, Wagner AJ, Kawai A, Tamura K, Shahir A, Van Tine BA, Martin-Broto J, Peterson PM, Wright J, Tap WD. Prospective Evaluation of Doxorubicin Cardiotoxicity in Patients with Advanced Soft-tissue Sarcoma Treated in the ANNOUNCE Phase III Randomized Trial. Clin Cancer Res. 2021 Jul 15;27(14):3861-3866. doi: 10.1158/1078-0432.CCR-20-4592. Epub 2021 Feb 25. PMID 33632930
- [Derived] Tap WD, Wagner AJ, Schoffski P, Martin-Broto J, Krarup-Hansen A, Ganjoo KN, Yen CC, Abdul Razak AR, Spira A, Kawai A, Le Cesne A, Van Tine BA, Naito Y, Park SH, Fedenko A, Papai Z, Soldatenkova V, Shahir A, Mo G, Wright J, Jones RL; ANNOUNCE Investigators. Effect of Doxorubicin Plus Olaratumab vs Doxorubicin Plus Placebo on Survival in Patients With Advanced Soft Tissue Sarcomas: The ANNOUNCE Randomized Clinical Trial. JAMA. 2020 Apr 7;323(13):1266-1276. doi: 10.1001/jama.2020.1707. PMID 32259228
- [Derived] Tobias A, O'brien MP, Agulnik M. Olaratumab for advanced soft tissue sarcoma. Expert Rev Clin Pharmacol. 2017 Jul;10(7):699-705. doi: 10.1080/17512433.2017.1324295. Epub 2017 May 5. PMID 28447475
- See also: A Study of Doxorubicin Plus Olaratumab (LY3012207) in Participants With Advanced or Metastatic Soft Tissue Sarcoma — https://trials.lillytrialguide.com/en-US/trial/1kxWhoB2GsgKesCo08Gmim

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers include participants who died in the study.
Groups:
- Doxorubicin + Olaratumab: 75 milligrams per meter squared (mg/m^2) doxorubicin administered intravenously (IV) on day 1 of each 21 day cycle up to 8 cycles plus 20 milligrams per kilogram (mg/kg) dose of olaratumab administered IV on day 1 and day 8 of cycle 1 and 15 mg/kg olaratumab administered IV on day 1 and day 8 of cycles 2-8. 15 mg/kg olaratumab administered IV on day 1 and day 8 of each subsequent 21 day cycle thereafter until documented progressive disease (PD) or discontinuation for any other reason.
- Doxorubicin + Placebo: 75 mg/m^2 doxorubicin administered IV on day 1 of each 21 day cycle up to 8 cycles plus placebo (equivalent volume) administered IV on day 1 and day 8 for 8 cycles. Placebo (equivalent volume) administered on days 1 and 8 of each subsequent 21 day cycle thereafter until PD or discontinuation for any other reason.
Period: Overall Study
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Started | 258 | 251
Received at Least One Dose of Study Drug | 257 | 249
Completed | 242 | 227
Not Completed | 16 | 24
Not completed — Withdrawal by Subject | 13 | 16
Not completed — Lost to Follow-up | 3 | 4
Not completed — Sponsor Decision | 0 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Doxorubicin + Olaratumab: 75 milligrams per meter squared (mg/m^2) doxorubicin administered intravenously (IV) on day 1 of each 21 day cycle for 8 cycles plus 20 milligrams per kilogram (mg/kg) dose of olaratumab administered IV on day 1 and day 8 of cycle 1 and 15 mg/kg olaratumab administered IV on day 1 and day 8 of cycles 2-8. Beginning with cycle 9, 15 mg/kg olaratumab administered IV on day 1 and day 8 of each subsequent 21 day cycle until documented progressive disease (PD) or discontinuation for any other reason.
- Doxorubicin + Placebo: 75 mg/m^2 doxorubicin administered IV on day 1 of each 21 day cycle for 8 cycles plus placebo (equivalent volume) administered IV on day 1 and day 8 for 8 cycles. Beginning with cycle 9, placebo (equivalent volume) administered on days 1 and 8 of each subsequent 21 day cycle until PD or discontinuation for any other reason.
- Total: Total of all reporting groups
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo | Total
Number analyzed (Participants) | 258 | 251 | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (12.4) | 57.1 (11.6) | 56.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 152 | 296
  Male | 114 | 99 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 29 | 55
  Not Hispanic or Latino | 209 | 199 | 408
  Unknown or Not Reported | 23 | 23 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 50 | 48 | 98
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 2 | 14
  White | 186 | 193 | 379
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69 | 73 | 142
  Russia | 7 | 8 | 15
  Austria | 3 | 0 | 3
  South Korea | 15 | 13 | 28
  Netherlands | 8 | 6 | 14
  Sweden | 4 | 3 | 7
  Brazil | 2 | 0 | 2
  Poland | 3 | 2 | 5
  France | 17 | 18 | 35
  Argentina | 3 | 4 | 7
  Hungary | 9 | 11 | 20
  Japan | 23 | 22 | 45
  United Kingdom | 10 | 16 | 26
  Switzerland | 4 | 2 | 6
  Spain | 13 | 21 | 34
  Canada | 12 | 6 | 18
  Belgium | 11 | 10 | 21
  Finland | 4 | 2 | 6
  Taiwan | 6 | 7 | 13
  Denmark | 10 | 2 | 12
  Italy | 5 | 4 | 9
  Mexico | 7 | 6 | 13
  Israel | 6 | 5 | 11
  Australia | 0 | 1 | 1
  Germany | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization to the date of death due to any cause. For each participant, prior to data analysis, a reasonable effort was made to obtain the most up-to-date status (date of death or last date known to be alive). For any participant not known to have died as of the data cutoff date, OS was censored at the date the participant was last known to be alive. For any participant who withdrew consent for survival follow-up, OS was censored at the last date for which the participant provided consent for follow-up contact. The Kaplan-Meier method was used to estimate median parameters.
Time Frame: Randomization to Date of Death Due to Any Cause (Up to 35.8 Months)
Population: All randomized participants. Censored participants in Doxorubicin + Olaratumab arm = 87 and Doxorubicin + Placebo arm = 91
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Number analyzed (Participants) | 258 | 251
Months | 20.37 [17.84 to 22.90] | 19.75 [16.49 to 23.75]
Statistical Analysis 1: Comparison: Doxorubicin + Olaratumab vs Doxorubicin + Placebo; Test type: Superiority; p = 0.6945, Log Rank; Stratified; Hazard Ratio (HR) = 1.047, 95% CI 2-sided [0.841 to 1.303]

2. Primary Outcome: Overall Survival (OS) Leiomyosarcoma (LMS)
Description: as for outcome 1
Time Frame: Randomization to Date of Death Due to Any Cause (Up to 35.8 Months)
Population: All randomized participants with LMS. Censored participants in Doxorubicin + Olaratumab arm = 42 and Doxorubicin + Placebo arm = 40.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Number analyzed (Participants) | 119 | 115
Months | 21.55 [18.63 to 27.63] | 21.88 [17.54 to 25.07]
Statistical Analysis 1: Comparison: Doxorubicin + Olaratumab vs Doxorubicin + Placebo; Test type: Superiority; p = 0.7618, Log Rank; Stratified; Hazard Ratio (HR) = 0.951, 95% CI 2-sided [0.690 to 1.312]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined by (Response Evaluation Criteria In Solid Tumors RECIST v.1.1) as the time from the date of randomization to the first date of radiologic disease progression or death due to any cause. Progressive Disease (PD) is at least 20% increase in sum of diameters of target lesions, with reference being the smallest sum on study and plus absolute increase of at least 5 millimeter (mm), or unequivocal progression of non-target lesions, or 1 or more new lesions. Censoring for death or PD due to increase sum of target lesions is defined for each participant as the time from the date of randomization to the first date of radiographic documentation of 1 or more lesions. Censoring for death without progression is defined as the date of death if there is no prior or concurrent radiologic disease progression.
Time Frame: Randomization to Objective Progression or Death Due to Any Cause (Up to 35.8 Months)
Population: All randomized participants. Censored participants in the Doxorubicin + Olaratumab arm = 39 and the Doxorubicin + Placebo arm =34.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Number analyzed (Participants) | 258 | 251
Months | 5.42 [4.11 to 6.70] | 6.77 [5.49 to 8.08]
Statistical Analysis 1: Comparison: Doxorubicin + Olaratumab vs Doxorubicin + Placebo; Test type: Superiority; p = 0.0422, Log Rank; Stratified; Hazard Ratio (HR) = 1.231, 95% CI 2-sided [1.009 to 1.502]

4. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR): Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving a best overall response of complete response (CR) + partial response (PR). CR is the disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized. Best overall response is classified based on the overall responses assessed by study investigators according to RECIST v1.1.
Time Frame: Randomization to Objective Disease Progression or Death Due to Any Cause (Up to 35.8 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Number analyzed (Participants) | 258 | 251
percentage of participants | 14.0 [9.7 to 18.2] | 18.3 [13.5 to 23.1]

5. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR, PR, or Stable Disease (SD): Disease Control Rate (DCR)
Description: DCR was defined as the percentage of randomized participants achieving a best overall response of CR, PR, or SD per RECIST v.1.1. CR is the disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized. PD is at least 20% increase in sum of diameters of target lesions, with reference being the smallest sum on study and plus absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Randomization to Objective Disease Progression or Death Due to Any Cause (Up to 35.5 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Number analyzed (Participants) | 258 | 251
percentage of participants | 67.4 [61.7 to 73.2] | 75.7 [70.4 to 81.0]

6. Secondary Outcome: Time to First Worsening on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Scores
Description: Time to first worsening was calculated as the time from the first study drug dose to the first observation of worsening according to the EORTC QLQ-C30 Scoring Manual (Fayers et al. 2001). The EORTC QLQ-C30 self-reported general cancer instrument consists of 30 total items covered by 1 of 3 dimensions (1 global health status/QoL total score, 5 functional subscales [physical, role, cognitive, emotional, and social]), and 9 symptom subscales [fatigue/nausea/vomiting/pain/dyspnea/insomnia/appetite loss/constipation/diarrhea]). There are 28 questions answered on a 4-point scale where 1=Not at all (best) to 4=Very Much (worst) and 2 questions answered on a 7-point scale where 1=Very poor (worst) to 7= Excellent (best). A linear transformation was used to obtain total score ranging from 0 to 100 where "worsening" was defined as an increase of at least 10 points for the symptom scales or a decrease of at least 10 points for the functional scales and the global health status/QoL scale.
Time Frame: Randomization (Cycle 1) through Follow-up (Up to 35.8 Months)
Population: All randomized participants who completed at least 1 baseline assessment and at least 1 subsequent assessment during the study period.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Number analyzed (Participants) | 258 | 251
Months
  Global Health Status/QoL: number analyzed (Participants) | 201 | 197
  Global Health Status/QoL | 1.45 [1.41 to 2.10] | 1.84 [1.45 to 2.79]
  Role Functional Scale: number analyzed (Participants) | 202 | 190
  Role Functional Scale | 1.41 [0.99 to 1.48] | 1.41 [0.95 to 2.00]
  Physical Functional Scale: number analyzed (Participants) | 205 | 209
  Physical Functional Scale | 1.81 [1.45 to 2.14] | 2.79 [2.07 to 3.48]
  Emotional Functional Scale: number analyzed (Participants) | 168 | 171
  Emotional Functional Scale | 3.48 [2.50 to 4.37] | 2.83 [2.14 to 4.34]
  Cognitive Functional Scale: number analyzed (Participants) | 170 | 167
  Cognitive Functional Scale | 1.64 [1.41 to 2.14] | 1.45 [1.41 to 2.07]
  Social Functional Scale: number analyzed (Participants) | 189 | 171
  Social Functional Scale | 1.45 [1.38 to 1.64] | 1.41 [1.35 to 1.45]
  Fatigue Symptom Scale: number analyzed (Participants) | 210 | 204
  Fatigue Symptom Scale | 0.92 [0.76 to 1.25] | 0.89 [0.76 to 1.38]
  Nausea and Vomiting Symptom Scale: number analyzed (Participants) | 182 | 173
  Nausea and Vomiting Symptom Scale | 1.45 [1.41 to 1.64] | 1.41 [0.95 to 1.45]
  Pain Symptom Scale: number analyzed (Participants) | 185 | 183
  Pain Symptom Scale | 1.64 [1.41 to 2.10] | 2.10 [1.45 to 2.76]
  Dyspnea Symptom Scale: number analyzed (Participants) | 158 | 160
  Dyspnea Symptom Scale | 2.10 [1.45 to 2.76] | 2.07 [1.45 to 2.79]
  Insomnia Symptom Scale: number analyzed (Participants) | 151 | 160
  Insomnia Symptom Scale | 2.10 [1.45 to 2.79] | 1.58 [1.41 to 2.33]
  Appetite Loss Symptom Scale: number analyzed (Participants) | 182 | 170
  Appetite Loss Symptom Scale | 1.48 [1.45 to 2.04] | 1.64 [1.41 to 2.14]
  Financial Difficulties Scale: number analyzed (Participants) | 132 | 105
  Financial Difficulties Scale | 1.48 [1.41 to 2.14] | 1.45 [1.41 to 2.10]
  Constipation Symptom Scale: number analyzed (Participants) | 169 | 157
  Constipation Symptom Scale | 1.64 [1.41 to 2.10] | 1.41 [1.41 to 2.10]
  Diarrhea Symptom Scale: number analyzed (Participants) | 157 | 148
  Diarrhea Symptom Scale | 2.07 [1.45 to 2.79] | 2.79 [2.10 to 3.52]

7. Secondary Outcome: Change From Baseline to Maximum Improvement in Health Status Index Score on the EuroQol 5-Dimension 5-Level (EQ-5D-5L)
Description: The EQ-5D-5L is a standardized measure of health status used to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L consists of a descriptive system of the respondent's health which comprises the following 5 dimensions: (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Health status was calculated from a set of item weights to derive a score of 0 to 1, with 1 representing the best health status. United Kingdom (UK) weights were applied. The analysis includes all cycles for which at least 25% of participants in each arm have an assessment. For each participant a change from baseline was calculated for every post-baseline assessment by subtracting the baseline assessment result from the current assessment result. Maximum improvement (over baseline) was determined from the set of all post-baseline change scores.
Time Frame: Randomization through Follow-up (Up to 35.8 Months)
Population: All randomized participants who had a baseline and a post-baseline measurement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Number analyzed (Participants) | 221 | 219
score on a scale | -0.163 (0.236) | -0.171 (0.235)

8. Secondary Outcome: Time to First Worsening of the Brief Pain Inventory Short Form Modified (mBPI-sf) "Worst Pain Score"
Description: Time to first worsening of the brief pain inventory short form modified (mBPI-sf) "worst pain score" was defined as the time from the date of the first study drug dose (baseline date) to the first date of a "worst pain" score increase of greater than or equal to (≥) 2 points from baseline. The mBPI-sf is an 11-item instrument used as a multiple-item measure of cancer pain intensity ranging from 0 (no pain or does not interfere) and ranged through 10 (pain as bad as you can imagine or completely interferes).
Time Frame: Randomization through Follow-up (Up to 34.5 Months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Number analyzed (Participants) | 211 | 206
Months | 7.66 [6.01 to 9.63] | 8.08 [6.18 to 11.07]

9. Secondary Outcome: Duration of Overall Response (DoR)
Description: The duration of overall response was defined for each participant with a best response of CR or PR and measured from the time measurement criteria are first met for CR or PR (whichever is first recorded) until the first date that disease is recurrent or objective disease progression or death due to any cause is observed (taking as reference for PD the smallest measurements recorded on study).
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up to 33.4 Months)
Population: All randomized participants who have evaluable DoR data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Number analyzed (Participants) | 36 | 46
Months | 8.31 [6.87 to 12.35] | 4.80 [3.65 to 6.83]
Statistical Analysis 1: Comparison: Doxorubicin + Olaratumab vs Doxorubicin + Placebo; Test type: Superiority; p = 0.0934, Log Rank; Stratified; Hazard Ratio (HR) = 0.616, 95% CI 2-sided [0.347 to 1.093]

10. Secondary Outcome: Duration of Disease Control (DDC)
Description: Duration of disease control was defined for each participant with a best response of CR, PR, or stable disease (SD) as the time from randomization to the first date of disease progression or death due to any cause.
Time Frame: Date of CR, PR, or SD to Objective Disease Progression or Death Due to Any Cause (Up to 35.8 Months)
Population: All randomized participants who had evaluable DDC data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
Number analyzed (Participants) | 174 | 190
Months | 8.28 [6.93 to 9.72] | 8.34 [8.08 to 9.46]
Statistical Analysis 1: Comparison: Doxorubicin + Olaratumab vs Doxorubicin + Placebo; Test type: Superiority; p = 0.3347, Log Rank; Stratified; Hazard Ratio (HR) = 1.123, 95% CI 2-sided [0.892 to 1.413]

11. Secondary Outcome: Pharmacokinetics (PK) Clearance of Olaratumab Mean Parameter Estimate
Description: The PK systemic clearance parameter estimates from the current analysis are listed together with the population PK model estimates.
Time Frame: Cycle 1- 9: Day 1 and 8, Predose, 5 minutes Post dose and then every other cycle and follow-up (30 Days)
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (95% Confidence Interval); unit: Liter/hour (L/h)
Arm/Group | Doxorubicin + Olaratumab
Number analyzed (Participants) | 258
Liter/hour (L/h) | 0.0195 [0.0189 to 0.0203]

12. Secondary Outcome: PK: Volume of Distribution at Steady State (Vss) of Olaratumab: Mean Parameter Estimate
Description: The PK parameter estimates from the current analysis are listed together with the population PK model estimates. The Vss is the sum of central volume of distribution (V1) + peripheral volume of distribution (V2).
Time Frame: Cycle 1- 9: Day 1 and 8; Predose, 5 Minutes Post dose and then every other cycle and follow-up (30 Days)
Population: All randomized participants who had received at least one dose of study drug and had evaluable PK data.
Measure: Mean (95% Confidence Interval); unit: Liter (L)
Arm/Group | Doxorubicin + Olaratumab
Number analyzed (Participants) | 258
Liter (L) | 5.72 [5.28 to 6.17]

ADVERSE EVENTS:
Time Frame: Baseline Up To 41 Months
Description: All participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly. Based on the planned safety analysis, adverse event analysis was planned as per the treatments the participants received.
Arm/Group | Doxorubicin + Olaratumab | Doxorubicin + Placebo
All-Cause Mortality (participants affected / at risk) | 170/257 | 158/249
Serious Adverse Events (participants affected / at risk) | 105/257 | 89/249
Other Adverse Events (participants affected / at risk) | 248/257 | 244/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Doxorubicin + Olaratumab (N=257) | Doxorubicin + Placebo (N=249)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 34 (37) | 33 (37)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 8 (10) | 8 (8)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (5)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (3)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 7 (7)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (6) | 4 (7)
Platelet count decreased (Investigations) | 2 (2) | 2 (2)
Troponin increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 2 (3) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Sciatic nerve neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar artery dissection (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/144 (0) | 1/151 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin + Olaratumab (N=257) | Doxorubicin + Placebo (N=249)
Anaemia (Blood and lymphatic system disorders) | 115 (169) | 121 (230)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (13) | 9 (12)
Leukopenia (Blood and lymphatic system disorders) | 14 (36) | 11 (23)
Neutropenia (Blood and lymphatic system disorders) | 59 (131) | 59 (121)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (29) | 19 (35)
Abdominal pain (Gastrointestinal disorders) | 31 (43) | 44 (55)
Abdominal pain upper (Gastrointestinal disorders) | 17 (23) | 20 (23)
Constipation (Gastrointestinal disorders) | 86 (122) | 94 (144)
Diarrhoea (Gastrointestinal disorders) | 79 (123) | 76 (118)
Dry mouth (Gastrointestinal disorders) | 22 (23) | 19 (21)
Dyspepsia (Gastrointestinal disorders) | 28 (33) | 29 (34)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 (17) | 18 (19)
Nausea (Gastrointestinal disorders) | 154 (293) | 171 (369)
Stomatitis (Gastrointestinal disorders) | 79 (134) | 93 (167)
Vomiting (Gastrointestinal disorders) | 62 (78) | 70 (128)
Asthenia (General disorders) | 24 (42) | 30 (66)
Fatigue (General disorders) | 129 (181) | 133 (211)
Malaise (General disorders) | 11 (13) | 15 (20)
Oedema peripheral (General disorders) | 37 (44) | 25 (39)
Pyrexia (General disorders) | 50 (65) | 42 (61)
Nasopharyngitis (Infections and infestations) | 10 (12) | 16 (17)
Rhinitis (Infections and infestations) | 6 (6) | 13 (16)
Upper respiratory tract infection (Infections and infestations) | 25 (31) | 25 (30)
Urinary tract infection (Infections and infestations) | 20 (29) | 23 (28)
Alanine aminotransferase increased (Investigations) | 20 (29) | 21 (33)
Aspartate aminotransferase increased (Investigations) | 11 (12) | 20 (28)
Gamma-glutamyltransferase increased (Investigations) | 21 (25) | 19 (25)
Lymphocyte count decreased (Investigations) | 17 (47) | 17 (39)
Neutrophil count decreased (Investigations) | 92 (205) | 90 (256)
Platelet count decreased (Investigations) | 47 (122) | 46 (140)
Weight decreased (Investigations) | 25 (26) | 23 (25)
White blood cell count decreased (Investigations) | 68 (177) | 69 (181)
Decreased appetite (Metabolism and nutrition disorders) | 74 (108) | 93 (131)
Dehydration (Metabolism and nutrition disorders) | 18 (24) | 9 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (21) | 10 (14)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (18) | 14 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (40) | 22 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 35 (48) | 31 (38)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 (25) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (20) | 12 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 (37) | 27 (40)
Dizziness (Nervous system disorders) | 27 (44) | 35 (49)
Dysgeusia (Nervous system disorders) | 42 (50) | 47 (57)
Headache (Nervous system disorders) | 43 (61) | 42 (56)
Paraesthesia (Nervous system disorders) | 12 (15) | 16 (17)
Anxiety (Psychiatric disorders) | 17 (21) | 16 (17)
Insomnia (Psychiatric disorders) | 25 (29) | 34 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (54) | 66 (81)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 (53) | 39 (48)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 19 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 113 (116) | 127 (132)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (15) | 11 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (16) | 23 (26)
Rash (Skin and subcutaneous tissue disorders) | 13 (16) | 18 (20)
Hypertension (Vascular disorders) | 19 (23) | 24 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol: Study Protocol (2015-01-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT02451943/Prot_000.pdf
  • Study Protocol: Study Protocol (d) (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT02451943/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT02451943/SAP_002.pdf